CLINICAL TRIAL: NCT03031080
Title: The Effectiveness of Night Splinting After Collagenase Injection for Dupuytren's Contracture
Brief Title: BOND Study: the Benefit Of Night Splinting in Dupuytrens'
Acronym: BOND
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Intervention (Xiapex) was removed from the market
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 5396
Record Dates: First submitted 2017-01-23; First posted 2017-01-25 (Estimated); Last update posted 2021-09-27 (Actual); Status verified 2018-04

CONDITIONS: Dupuytren Contracture
Keywords: Collagenase, Night-splinting, Dupuytrens, Contracture
MeSH Terms: conditions — Dupuytren Contracture; Contracture

STUDY DESIGN:
Intervention Model Description: Randomised Controlled Trial - Block Randomisation
Who Masked: Investigator, Outcomes Assessor
Masking Description: Initial heath-care provider and participant are not masked as would be impossible to do so. Outcome assessor (a different health care provider) and investigators will be masked as to whether the patient is in the splinted or unsplinted cohort.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Splinted (Active Comparator): Patients will be given Thermoplastic Hand Splint to wear overnight for 12 weeks.
  Interventions: Device: Thermoplastic Hand Splint
- Un-Splinted (No Intervention): Patients will not wear a night splint

INTERVENTIONS:
Device: Thermoplastic Hand Splint — Thermoplastic Night splint created and moulded to the individual patients hand in-house using generic thermoplastic.
  Arms: Splinted

SUMMARY:
The BOND study is a prospective, randomised single blinded controlled trial to assess the effect of night splinting in patients who have had collagenase injection and manipulation therapy for Dupuytren's Contracture.

DETAILED DESCRIPTION:
This trial will assess the effectiveness of night splinting in Dupuytrens' contracture on functional and quality of life outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Single digit contractures greater than 30 degrees
2. No prior surgery for their contractures.
3. Successful collagenase and manipulation therapy (contracture reduced to within 10 degrees of full extension).

Exclusion Criteria:

1. Multiple digit contractures
2. Prior surgery for their contractures.
3. Failure of collagenase and manipulation therapy (contracture not reduced to within 10 degrees of full extension).
4. Inability to consent to treatment.

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2018-12-31 (Estimated); Study Completion 2019-06-30 (Estimated)

PRIMARY OUTCOMES:
Range of motion | At 0 weeks, 12 weeks and 52 weeks
  To assess change in range of motion measured in degrees between pre-treatment, immediately post-treatment, 12 weeks post-treatment and 12 months post-treatment

SECONDARY OUTCOMES:
PEM Questionnaire | At 0 weeks, 12 weeks and 52 weeks
  Patient Evaluation Measure to give disability score
URAM Questionnaire | At 0 weeks, 12 weeks and 52 weeks
  Hand specific outcome questionnaire to assess quality of life outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Graham Cheung, MBBCh FRCS, Principal Investigator — Consultant Hand Surgeon
Locations (1):
- Royal Liverpool & Broadgreen University Hospitals NHS Trust, Liverpool, Merseyside, United Kingdom

IPD SHARING:
Plan to Share IPD: No